CLINICAL TRIAL: NCT00829075
Title: A Prospective, Randomized, Controlled Trial Comparing Three Different Gonadotrophin Regimens in Oocyte Donors: Ovarian Response and IVF Outcome
Brief Title: Impact of Three Different Gonadotrophin Regimes on Egg Donation Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Marco Melo, IVI Valencia
Other Study IDs: VLC-MM-0501-37
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Ovarian Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Experimental): only r-FSH TREATMENT
  Interventions: Drug: r-FSH
- II (Experimental): only HP-hMG TREATMENT
  Interventions: Drug: HP-hMG
- III (Experimental): r-FSH plus HP-hMG TREATMENT
  Interventions: Drug: r-FSH plus HP-hMG

INTERVENTIONS:
Drug: r-FSH
  Arms: I
Drug: HP-hMG
  Arms: II
Drug: r-FSH plus HP-hMG
  Arms: III

SUMMARY:
Exploratory study assessing the effect of three gonadotrophin protocols on Controlled Ovarian Stimulation (COS) parameters and IVF outcome in oocyte donors undergoing GnRH analogue (long protocol). 1,028 donors were randomized in three groups: Group I (n= 346) only r-FSH, Group II (n= 333) only HP-hMG and Group III (n= 349) r-FSH plus HP-hMG. IVF outcome of 1,059 oocyte recipients was compared.

ELIGIBILITY:
Inclusion Criteria:

* healthy women 18-34 years of age
* regular menstrual cycles
* no family history of hereditary or chromosomal diseases
* normal karyotype
* BMI 18-29 Kg/m2
* negative screening for sexually transmitted diseases

Exclusion Criteria:

* women with PCOS were not included in this study

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The aim of this study was to verify whether different gonadotrophin regimes could affect controlled ovarian stimulation (COS) parameters and IVF outcome in an egg donation program. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marco Melo, MDPhD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Spain